CLINICAL TRIAL: NCT02417025
Title: Do You Really Expect Me to Get MST Care in a VA Where Everyone is Male? Innovative Delivery of Evidence Based Psychotherapy to Women With Military Sexual Trauma (MST)
Brief Title: Innovative Delivery of Evidence Based Psychotherapy to Women With Military Sexual Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Charleston Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00034989
Record Dates: First submitted 2014-12-15; First posted 2015-04-15 (Estimated); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: PTSD; Stress Disorders, Post - Traumatic; Anxiety Disorders; Mental Disorders; Stress Disorders, Traumatic
Keywords: Military; Health Service Delivery; Telepsychology; Prolonged Exposure; Off-duty Activity of Military Personnel
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Combat Disorders; Anxiety Disorders; Mental Disorders; Stress Disorders, Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PE-HBT (Experimental): Prolonged Exposure via home-based telehealth (i.e., completed using videoconferencing technology)
  Interventions: Behavioral: PE
- PE-SD (Active Comparator): Prolonged Exposure via standard delivery (i.e., completed in person at the therapist's office)
  Interventions: Behavioral: PE

INTERVENTIONS:
Behavioral: PE — Prolonged Exposure

SUMMARY:
The purpose of this study is to determine whether a scientifically validated treatment for Posttraumatic Stress Disorder (PTSD) called Prolonged Exposure (PE) can be delivered effectively to Veterans with Military Sexual Trauma (MST) related PTSD using videoconferencing technology, which allows a therapist and patient who are not in the same room as one another to communicate. The investigators are interested in learning if this form of mental health service delivery is an acceptable alternative to traditional face-to-face therapy delivered with the therapist in the same room as the patient. This study is being conducted at the Charleston VA Medical Center and surrounding Community-Based Outpatient Clinics (CBOCs), and will involve approximately 100 female participants.

DETAILED DESCRIPTION:
The purpose of this project is to test, using mixed qualitative and quantitative assessment strategies, the efficacy of PE delivered via home-based telehealth (PE-HBT) versus PE delivered via standard service delivery (PE-SD) using a randomized, between groups, repeated measures design.

Objective 1: To compare, at post, 3 and 6-month follow-up, whether PE-HBT is superior to PE-SD across critical clinical and quality of life outcomes (i.e., PTSD, depression, quality of life) due to increased PE 'dosing' that results from improved session attendance and reduced attrition.

Hypothesis 1: In intent-to-treat analyses, PE-HBT will be more effective than PE-SD at improving clinical and quality of life outcomes at post, 3, and 6-month follow-up; improvement will correlate with session attendance, which will be higher in PE-HBT.

Objective 2: To compare at post-intervention whether PE-HBT is superior to PE-SD across critical process outcomes (e.g., session attendance, satisfaction, and treatment adherence).

Hypothesis 2: PE-HBT will yield better process outcomes than PE-SD post-intervention.

Exploratory Aims: (1) To determine if treatment adherence and other process variables mediate the relationship between treatment condition and clinical and quality of life outcomes as noted in Objective 1; and (2) To use qualitative interviewing methods to obtain data on Veterans' reactions, preferences, difficulties, and suggestions for MST services.

ELIGIBILITY:
Inclusion Criteria:

1. MST-related index event
2. Diagnosis of PTSD-related MST
3. Female

Exclusion Criteria:

1. Having a household member of spouse who is already enrolled in the study
2. Active psychosis or dementia
3. Suicidal and/or homicidal ideation with clear intent
4. Current substance dependence
5. Concurrent enrollment in another clinical trial for PTSD or depression
6. Unwilling to make regular appointments (note that if the participant has medical/transportation barriers that render her unable to make set appointments, this is not grounds for exclusion).

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2014-08; Primary Completion 2019-11-29 (Actual); Study Completion 2019-11-29 (Actual)

PRIMARY OUTCOMES:
Number of Participants Receiving Prolonged Exposure Treatment via Telemedicine with significantly decreased PTSD symptoms Compared to Number of Participants Receiving Prolonged Exposure Treatment with Standard In-Person Delivery | 36 weeks

SECONDARY OUTCOMES:
Veteran (VR) Short Form (SF) -12 Health Survey (VR-12) | Baseline
  The VR-12 is short measure designed to assess participants' views on their current health, how they are feeling at this time point, and how well they are able to do their usual activities. It also asks questions regarding how daily activities are/have been hindered by problems with their physical health.
Veteran (VR) Short Form (SF) -12 Health Survey (VR-12) | 13 weeks
  The VR-12 is short measure designed to assess participants' views on their current health, how they are feeling at this time point, and how well they are able to do their usual activities. It also asks questions regarding how daily activities are/have been hindered by problems with their physical health.
Veteran (VR) Short Form (SF) -12 Health Survey (VR-12) | 24 weeks
  The VR-12 is short measure designed to assess participants' views on their current health, how they are feeling at this time point, and how well they are able to do their usual activities. It also asks questions regarding how daily activities are/have been hindered by problems with their physical health.
Veteran (VR) Short Form (SF) -12 Health Survey (VR-12) | 36 weeks
  The VR-12 is short measure designed to assess participants' views on their current health, how they are feeling at this time point, and how well they are able to do their usual activities. It also asks questions regarding how daily activities are/have been hindered by problems with their physical health.
Index of Functional Impairment (IFI) | Baseline
  The Index of Functional Impairment (IFI) is a self-report inventory of functional impairment. Patients rate their level of functioning across multiple psychosocial domains including romantic relationships, employment, and educational achievement.
Index of Functional Impairment (IFI) | 13 weeks
  The Index of Functional Impairment (IFI) is a self-report inventory of functional impairment. Patients rate their level of functioning across multiple psychosocial domains including romantic relationships, employment, and educational achievement.
Index of Functional Impairment (IFI) | 24 weeks
  The Index of Functional Impairment (IFI) is a self-report inventory of functional impairment. Patients rate their level of functioning across multiple psychosocial domains including romantic relationships, employment, and educational achievement.
Index of Functional Impairment (IFI) | 36 weeks
  The Index of Functional Impairment (IFI) is a self-report inventory of functional impairment. Patients rate their level of functioning across multiple psychosocial domains including romantic relationships, employment, and educational achievement.
Treatment Credibility Questionnaire | 13 weeks
  This questionnaire is used to assess for differences in outcome expectancy using treatment credibility scales. The questionnaire asks how the participant feels about the current treatment she is receiving, how logical it seems, how likely she would be to recommend it to a friend, and how successful she believes it is in decreasing different symptoms of PTSD, such as fear.
Charleston Psychiatric Outpatient Satisfaction Scale (CPOSS) | 13 weeks
  The CPOSS is a 16-item questionnaire that assesses the participant's attitudes about the Charleston VA facility, such as the quality of care she received at the hospital, the helpfulness of the secretary, clear and correct monthly documentation of problems in her medical record, etc.
Mini International Neuropsychiatric Interview (M.I.N.I.) | Baseline
  The MINI is a brief structured interview that assesses the criteria for DSM-V Axis I diagnoses. The MINI will be used to assess for a diagnosis of current depression, panic symptoms, generalized anxiety symptoms, eating disorders, psychotic symptoms and to screen for substance dependence.
Mini International Neuropsychiatric Interview (M.I.N.I.) | 36 weeks
  The MINI is a brief structured interview that assesses the criteria for DSM-V Axis I diagnoses. The MINI will be used to assess for a diagnosis of current depression, panic symptoms, generalized anxiety symptoms, eating disorders, psychotic symptoms and to screen for substance dependence.
Alcohol Use Disorder Identification Test (AUDIT) | Baseline
  The AUDIT is a 10-item measure that assesses the level of the participant's drinking. Questions include how many drinks a participant has during a day or on occasions, possible harmful consequences of drinking, and feelings of remorse about drinking.
Alcohol Use Disorder Identification Test (AUDIT) | 13 weeks
  The AUDIT is a 10-item measure that assesses the level of the participant's drinking. Questions include how many drinks a participant has during a day or on occasions, possible harmful consequences of drinking, and feelings of remorse about drinking.
Alcohol Use Disorder Identification Test (AUDIT) | 24 weeks
  The AUDIT is a 10-item measure that assesses the level of the participant's drinking. Questions include how many drinks a participant has during a day or on occasions, possible harmful consequences of drinking, and feelings of remorse about drinking.
Alcohol Use Disorder Identification Test (AUDIT) | 36 weeks
  The AUDIT is a 10-item measure that assesses the level of the participant's drinking. Questions include how many drinks a participant has during a day or on occasions, possible harmful consequences of drinking, and feelings of remorse about drinking.
Drug Abuse Screening Test (DAST-10) | Baseline
  The DAST-10 is a 10-item measure designed to assess for illegal drug use (not including alcohol) for the past month.
Drug Abuse Screening Test (DAST-10) | 13 weeks
  The DAST-10 is a 10-item measure designed to assess for illegal drug use (not including alcohol) for the past month.
Drug Abuse Screening Test (DAST-10) | 24 weeks
  The DAST-10 is a 10-item measure designed to assess for illegal drug use (not including alcohol) for the past month.
Drug Abuse Screening Test (DAST-10) | 36 weeks
  The DAST-10 is a 10-item measure designed to assess for illegal drug use (not including alcohol) for the past month.
Pittsburgh Sleep Quality Index (PSQI) | Baseline
  The PSQI is a 19-item commonly used and well validated self-report measure of sleep quality and disturbance. Scores on the PSQI range from 0 to 21, with rating of 5 or higher indicative of poor sleep quality.
Pittsburgh Sleep Quality Index (PSQI) | 13 weeks
  The PSQI is a 19-item commonly used and well validated self-report measure of sleep quality and disturbance. Scores on the PSQI range from 0 to 21, with rating of 5 or higher indicative of poor sleep quality.
Pittsburgh Sleep Quality Index (PSQI) | 24 weeks
  The PSQI is a 19-item commonly used and well validated self-report measure of sleep quality and disturbance. Scores on the PSQI range from 0 to 21, with rating of 5 or higher indicative of poor sleep quality.
Pittsburgh Sleep Quality Index (PSQI) | 36 weeks
  The PSQI is a 19-item commonly used and well validated self-report measure of sleep quality and disturbance. Scores on the PSQI range from 0 to 21, with rating of 5 or higher indicative of poor sleep quality.
Sexual Assault Related Mental Contamination Scale (SARA) | Baseline
  This abbreviated version of the 80-item SARA scale assesses the participant's perceptions of her sexual assault/rape.
Sexual Assault Related Mental Contamination Scale (SARA) | 13 weeks
  This abbreviated version of the 80-item SARA scale assesses the participant's perceptions of her sexual assault/rape.
Sexual Assault Related Mental Contamination Scale (SARA) | 24 weeks
  This abbreviated version of the 80-item SARA scale assesses the participant's perceptions of her sexual assault/rape.
Sexual Assault Related Mental Contamination Scale (SARA) | 36 weeks
  This abbreviated version of the 80-item SARA scale assesses the participant's perceptions of her sexual assault/rape.
Beck Depression Inventory - II (BDI-II) | Baseline
  Beck Depression Inventory-II is a 21 item measure of depressive severity with higher total scores indicative of more severe depression.
Beck Depression Inventory - II (BDI-II) | 13 weeks
  Beck Depression Inventory-II is a 21 item measure of depressive severity with higher total scores indicative of more severe depression.
Beck Depression Inventory - II (BDI-II) | 24 weeks
  Beck Depression Inventory-II is a 21 item measure of depressive severity with higher total scores indicative of more severe depression.
Beck Depression Inventory - II (BDI-II) | 36 weeks
  Beck Depression Inventory-II is a 21 item measure of depressive severity with higher total scores indicative of more severe depression.
PTSD Checklist, 5th Version (PCL-5) | Baseline
  The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. The PCL-5 has a variety of purposes, including, monitoring symptom change during and after treatment, screening individuals for PTSD, and making a provisional PTSD diagnosis. Description information provided by the National Center for PTSD.
PTSD Checklist, 5th Version (PCL-5) | 13 weeks
  The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. The PCL-5 has a variety of purposes, including, monitoring symptom change during and after treatment, screening individuals for PTSD, and making a provisional PTSD diagnosis. Description information provided by the National Center for PTSD.
PTSD Checklist, 5th Version (PCL-5) | 24 weeks
  The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. The PCL-5 has a variety of purposes, including, monitoring symptom change during and after treatment, screening individuals for PTSD, and making a provisional PTSD diagnosis. Description information provided by the National Center for PTSD.
PTSD Checklist, 5th Version (PCL-5) | 36 weeks
  The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. The PCL-5 has a variety of purposes, including, monitoring symptom change during and after treatment, screening individuals for PTSD, and making a provisional PTSD diagnosis. Description information provided by the National Center for PTSD.
Clinical Administrated PTSD Scale (CAPS) | Baseline
  The Clinician Administered PTSD (Posttraumatic stress disorder) Scale (CAPS) is a 30-item structured interview that corresponds to the Diagnostic and Statistical Manual of Mental Disorders, 5th Version (DSM-V) criteria for PTSD. The CAPS can be used to make a current (past month) or lifetime diagnosis of PTSD or to assesses symptoms over the past week.
Clinical Administrated PTSD Scale (CAPS) | 13 weeks
  The Clinician Administered PTSD (Posttraumatic stress disorder) Scale (CAPS) is a 30-item structured interview that corresponds to the Diagnostic and Statistical Manual of Mental Disorders, 5th Version (DSM-V) criteria for PTSD. The CAPS can be used to make a current (past month) or lifetime diagnosis of PTSD or to assesses symptoms over the past week.
Clinical Administrated PTSD Scale (CAPS) | 24 weeks
  The Clinician Administered PTSD (Posttraumatic stress disorder) Scale (CAPS) is a 30-item structured interview that corresponds to the Diagnostic and Statistical Manual of Mental Disorders, 5th Version (DSM-V) criteria for PTSD. The CAPS can be used to make a current (past month) or lifetime diagnosis of PTSD or to assesses symptoms over the past week.
Clinical Administrated PTSD Scale (CAPS) | 36 weeks
  The Clinician Administered PTSD (Posttraumatic stress disorder) Scale (CAPS) is a 30-item structured interview that corresponds to the Diagnostic and Statistical Manual of Mental Disorders, 5th Version (DSM-V) criteria for PTSD. The CAPS can be used to make a current (past month) or lifetime diagnosis of PTSD or to assesses symptoms over the past week.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald E Acierno, PhD, Principal Investigator — Ralph H. Johnson VA Medical Center
Locations (1):
- Ralph H. Johnson VAMC, Charleston, South Carolina, United States

REFERENCES:
- [Derived] Acierno R, Jaffe AE, Gilmore AK, Birks A, Denier C, Muzzy W, Lopez CM, Tuerk P, Grubaugh AL. A randomized clinical trial of in-person vs. home-based telemedicine delivery of Prolonged Exposure for PTSD in military sexual trauma survivors. J Anxiety Disord. 2021 Oct;83:102461. doi: 10.1016/j.janxdis.2021.102461. Epub 2021 Aug 8. PMID 34391978